CLINICAL TRIAL: NCT07122570
Title: Outcomes After Total Elbow Arthroplasty Using the Latitude Elbow Prosthesis: A 2-year Observational Study
Brief Title: Outcomes After Total Elbow Arthroplasty
Status: Completed | Type: Observational
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Latitude
Record Dates: First submitted 2022-07-14; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Elbow Disease
Keywords: arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will be an observational study involving patients from Wrightington hospital who underwent implantation of a Latitude elbow prosthesis a minimum of 2 years ago.

ELIGIBILITY:
Inclusion Criteria:

All patients who have undergone primary total elbow arthroplasty at Wrightington hospital between January 2014 and June 2018 with a Latitude total elbow prosthesis

Exclusion Criteria:

Patients who have undergone TEA with any elbow joint prosthesis other than the Latitude convertible total elbow joint prosthesis Patients whose TEA was not a primary procedure Patient not giving consent for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who had a Latitude elbow replacement for elbow arthritis
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Implant survival at 2 years post-surgery using a Kaplan-Meier estimate. | survival after surgical intervention
  standard statistical methods of Kaplan-Meier

SECONDARY OUTCOMES:
Oxford Shoulder Score | a single time point at 2 years or more after surgical intervention
  The Oxford Elbow Score has 12 items (questions) with 5 response options each. Each item response is scored 0 to 4, with 0 representing greater severity.
ELBEX | a single time point at 2 years or more after surgical intervention
  a pain section, which uses three 0-10 visual analogue scale scores to record the worst pain experienced from the elbow. also contains a function section, which lists 10 activities of daily living and asks the participant to rate the level of difficulty they experience with that activity using a series of 0-10 scales)
Quick DASH | a single time point at 2 years or more after surgical intervention
  QuickDASH only contains 11 items. It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms
ASES | a single time point at 2 years or more after surgical intervention
  divided into three sections: pain, function and satisfaction. The first section contains visual analogical scales (from 0 no pain to 10 worst pain ever) for pain evaluation. The second section contains questions relating to the function of the upper limbs

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Trail, Principal Investigator — Wrightington, Wigan & Leigh Teaching Hospital NHS Foundation Trust
Locations (1):
- Wrightington, Wigan & Leigh Teaching Hospitals NHS Foundation Trust, Wigan, United Kingdom